CLINICAL TRIAL: NCT03355573
Title: A Multicenter, Open-Label Extension Study to Evaluate the Long Term Safety and Efficacy of Bimekizumab in Subjects With Ankylosing Spondylitis
Brief Title: A Study to Evaluate the Long Term Safety and Efficacy of Bimekizumab in Subjects With Ankylosing Spondylitis
Acronym: BE AGILE 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS0009; 2017-001002-15 (EudraCT Number)
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Ankylosing Spondylitis
Keywords: Bimekizumab; Ankylosing Spondylitis; AS
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bimekizumab (Experimental): Subjects will receive bimekizumab up to 4 years.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab at a prespecified dose.
  Other Names: UCB4940

SUMMARY:
This is a study to assess the long term safety and tolerability of bimekizumab in subjects with ankylosing spondylitis

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the Investigator, the subject is expected to benefit from participation in an Open Label Extension (OLE) study
* Subject completed AS0008 without meeting any withdrawal criteria
* Female subjects must be postmenopausal, permanently sterilized or, if of childbearing potential, must be willing to use a highly effective method of contraception
* Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active

Exclusion Criteria:

* Female subjects who plan to become pregnant during the study or within 20 weeks following the last dose of investigational medicinal product (IMP). Male subjects who are planning a partner pregnancy during the study or within 20 weeks following the last dose
* Subjects with any current sign or symptom that may indicate a medically significant active infection (except for the common cold) or has had an infection requiring systemic antibiotics within 2 weeks of study entry
* Subjects who meet any withdrawal criteria in AS0008. For any subject with an ongoing Serious Adverse Event, or a history of serious infections (including hospitalizations) in the lead-in study, the Medical Monitor must be consulted prior to the subject's entry into AS0009

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (50):
- United States (3):
  - As0009 30, Sarasota, Florida
  - AS0009 1, Duncansville, Pennsylvania
  - AS0009 6, Dallas, Texas
- Bulgaria (4):
  - As0009 156, Dobrich
  - As0009 151, Plovdiv
  - As0009 155, Plovdiv
  - As0009 150, Rousse
- As0009 101, Québec, Canada
- Czechia (8):
  - As0009 205, Brno
  - As0009 207, Olomouc
  - As0009 208, Pardubice
  - As0009 201, Prague
  - As0009 202, Prague
  - As0009 211, Prague
  - As0009 210, Praha 11 Chodov
  - As0009 203, Zlín
- Germany (2):
  - As0009 304, Hamburg
  - As0009 301, Ratingen
- Hungary (3):
  - As0009 400, Budapest
  - As0009 403, Budapest
  - As0009 401, Veszprém
- Poland (13):
  - As0009 466, Bydgoszcz
  - As0009 453, Elblag
  - As0009 456, Elblag
  - As0009 455, Krakow
  - As0009 461, Lublin
  - As0009 467, Nowa Sól
  - As0009 451, Poznan
  - As0009 450, Torun
  - As0009 454, Warsaw
  - As0009 459, Warsaw
  - As0009 457, Wroclaw
  - As0009 460, Wroclaw
  - As0009 465, Wroclaw
- Russia (7):
  - As0009 601, Moscow
  - As0009 604, Moscow
  - As0009 607, Moscow
  - As0009 600, Saint Petersburg
  - As0009 606, Saint Petersburg
  - As0009 608, Saint Petersburg
  - As0009 610, Saint Petersburg
- Spain (3):
  - As0009 801, A Coruña
  - As0009 800, Córdoba
  - As0009 803, Santiago de Compostela
- Ukraine (6):
  - As0009 700, Kyiv
  - As0009 707, Kyiv
  - As0009 705, Ternopil
  - As0009 708, Uzhhorod
  - As0009 706, Vinnytsia
  - As0009 704, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baraliakos X, Deodhar A, Dougados M, Gensler LS, Molto A, Ramiro S, Kivitz AJ, Poddubnyy D, Oortgiesen M, Vaux T, Fleurinck C, Shepherd-Smith J, de la Loge C, de Peyrecave N, van der Heijde D. Safety and Efficacy of Bimekizumab in Patients With Active Ankylosing Spondylitis: Three-Year Results From a Phase IIb Randomized Controlled Trial and Its Open-Label Extension Study. Arthritis Rheumatol. 2022 Dec;74(12):1943-1958. doi: 10.1002/art.42282. Epub 2022 Nov 7. PMID 35829672
- [Result] Robinson PC, Machado PM, Haroon N, Gensler LS, Reveille JD, Taieb V, Vaux T, Fleurinck C, Oortgiesen M, de Peyrecave N, Deodhar A. Minimal Impact of the COVID-19 Pandemic on Disease Activity and Health-Related Quality of Life in Patients With Ankylosing Spondylitis Receiving Bimekizumab: Exploratory Analyses From a Phase 2b Open-Label Extension Study. ACR Open Rheumatol. 2022 Sep;4(9):819-824. doi: 10.1002/acr2.11486. Epub 2022 Jul 14. PMID 35833532
- [Result] Brown MA, Rudwaleit M, van Gaalen FA, Haroon N, Gensler LS, Fleurinck C, Marten A, Massow U, de Peyrecave N, Vaux T, White K, Deodhar A, van der Horst-Bruinsma I. Low uveitis rates in patients with axial spondyloarthritis treated with bimekizumab: pooled results from phase 2b/3 trials. Ann Rheum Dis. 2024 Nov 14;83(12):1722-1730. doi: 10.1136/ard-2024-225933. PMID 38977276
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794
- [Derived] Deodhar A, Navarro-Compan V, Poddubnyy D, Gensler LS, Ramiro S, Tomita T, Marzo-Ortega H, Fleurinck C, Vaux T, Massow U, de Peyrecave N, van der Heijde D, Baraliakos X. Long-term safety and sustained efficacy of bimekizumab in patients with ankylosing spondylitis (radiographic axial spondyloarthritis): 5-year results from BE AGILE (phase 2b) and its open-label extension. RMD Open. 2025 Jan 31;11(1):e005081. doi: 10.1136/rmdopen-2024-005081. PMID 39890205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in November 2017 and concluded in October 2022. Participants who completed AS0008 (NCT02963506) participated in this study.
Pre-assignment Details: The Participant Flow refers to the Safety Set.
Groups:
- Bimekizumab: Participants received bimekizumab 160 milligrams (mg) every 4 weeks (Q4W) up to 4 years.
Period: Overall Study
Arm/Group | Bimekizumab
Started | 255
Completed | 202
Not Completed | 53
Not completed — Withdrew consent due to refused treatment to AE latent tuberculosis | 1
Not completed — Sponsor's decision | 1
Not completed — Participant withdrew consent due to AEs | 1
Not completed — PI's decision | 2
Not completed — Withdrawal by Subject | 23
Not completed — Lost to Follow-up | 4
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event, non-fatal | 17
Not completed — Adverse Event, serious fatal | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set consisted of all participants in the enrolled set who received at least one dose of study medication in AS0009.
Groups:
- Bimekizumab: Participants received Bimekizumab 160 mg Q4W up to 4 years.
Arm/Group | Bimekizumab
Number analyzed (Participants) | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 245
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 217
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 253
  Other/Mixed | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 254

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Treatment emergent adverse events were defined as those events with onset date on or after the first administration of study medication in AS0009 and on or before 140 days after the final study medication administration.
Time Frame: From Entry Visit (Visit 1) until Safety Follow Up (up to Week 224)
Population: The Safety Set consisted of all participants in the enrolled set who received at least one dose of study medication in AS0009.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab
Number analyzed (Participants) | 255
percentage of participants | 92.9

2. Primary Outcome: Percentage of Participants With Serious Adverse Event (SAE) During the Study
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose: 1) Results in death 2) Is life-threatening 3) Requires in participant hospitalisation or prolongation of existing hospitalisation 4) Is a congenital anomaly or birth defect 5) Is an infection that requires treatment with parenteral antibiotics 6) Other important medical events which based on medical or scientific judgement may jeopardise the participants, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Entry Visit (Visit 1) until Safety Follow Up (up to Week 224)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab
Number analyzed (Participants) | 255
percentage of participants | 18.0

3. Secondary Outcome: Percentage of Participants Who Withdrew Due to an Treatment-emergent Adverse Event (TEAE) During the Study
Description: as for outcome 1
Time Frame: From Entry Visit (Visit 1) until Safety Follow Up (up to Week 224)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab
Number analyzed (Participants) | 255
percentage of participants | 6.7

4. Secondary Outcome: Percentage of Participants With Axial Spondyloarthritis International Society 40% Response Criteria (ASAS40) at Week 48 Calculated Relative to Baseline of AS0008
Description: The ASAS40 response was defined as relative improvements of at least 40% and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS), where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA) (score ranged from 0 (not active) to 10 (very active), Pain assessment (total spinal pain NRS score) (assessed on a scale of 0 (no pain) to 10 (severe pain)), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)) (score ranged from 0 (easy) to 10 (impossible)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) (score ranged from 0 (none) to 10 (very severe) and no worsening at all in the remaining domain. Participants for whom ASAS could not be derived due to missing data were counted as non-responders.
Time Frame: Baseline of AS0008, Week 48 (AS0009)
Population: The Full Analysis Set consisted of all enrolled participants who received at least 1 dose of the IMP and had a valid measurement for at least 1 efficacy variable at AS0009 study entry. Both Non-responder imputation and observed case analysis (imputation methods) have been reported in this outcome measure. Here, Number analyzed signifies those participants evaluable at specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab
Number analyzed (Participants) | 249
percentage of participants
  Non-responder imputation | 67.1
  Observed case: number analyzed (Participants) | 237
  Observed case | 70.5

5. Secondary Outcome: Percentage of Participants With Axial Spondyloarthritis International Society 20% Response Criteria (ASAS20) at Week 48 Calculated Relative to Baseline of AS0008
Description: The ASAS20 response was defined as relative improvements of at least 20% and absolute improvement of at least 1 unit on a 0 to 10 NRS, where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: PGADA (score ranged from 0 (not active) to 10 (very active), Pain assessment (total spinal pain NRS score) (assessed on a scale of 0 (no pain) to 10 (severe pain)), Function (BASFI) (score ranged from 0 (easy) to 10 (impossible)), Inflammation (mean of BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) (score ranged from 0 (none) to 10 (very severe) and no worsening at all in the remaining domain. Participants for whom ASAS could not be derived due to missing data were counted as non-responders.
Time Frame: Baseline of AS0008, Week 48 (AS0009)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab
Number analyzed (Participants) | 249
percentage of participants
  Non-responder imputation | 79.9
  Observed case: number analyzed (Participants) | 237
  Observed case | 84.0

6. Secondary Outcome: Change From Baseline of AS0008 in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score to Week 48
Description: BASDAI is a validated self-reported instrument, which consisted of 6 questions to measure the disease activity of ankylosing spondylitis (AS) from the participant's perspective. It measured the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration). Each question was rated using a numerical rating scale from 0 (none) to 10 (very severe), higher score=high disease activity. The BASDAI score was calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions 1 to 4. This score was then divided by 5. The total BASDAI score was ranged from 0=none to 10= very severe, where higher score indicated high disease activity. A negative value indicated improvement and a positive value indicated worsening.
Time Frame: Baseline of AS0008, Week 48 (AS0009)
Population: The Full Analysis Set consisted of all enrolled participants who received at least 1 dose of the IMP and had a valid measurement for at least 1 efficacy variable at AS0009 study entry.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Bimekizumab
Number analyzed (Participants) | 249
scores on a scale | -3.79 (0.13)

ADVERSE EVENTS:
Time Frame: From Entry Visit (Visit 1) until Safety Follow Up (up to Week 224)
Description: Treatment emergent adverse events were defined as those events with onset date on or after the first administration of study medication in AS0009 and on or before 140 days after the final study medication administration. The Safety Set consisted of all participants in the enrolled set who received at least one dose of study medication in AS0009.
Arm/Group | Bimekizumab
All-Cause Mortality (participants affected / at risk) | 2/255
Serious Adverse Events (participants affected / at risk) | 46/255
Other Adverse Events (participants affected / at risk) | 176/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab (N=255)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Endolymphatic hydrops (Ear and labyrinth disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Perirectal abscess (Infections and infestations) | 2 (2)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Corona virus infection (Infections and infestations) | 3 (3)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab (N=255)
Oral candidiasis (Infections and infestations) | 17 (21)
Bronchitis (Infections and infestations) | 21 (23)
Nasopharyngitis (Infections and infestations) | 46 (65)
Upper respiratory tract infection (Infections and infestations) | 33 (48)
Pharyngitis (Infections and infestations) | 18 (24)
Sinusitis (Infections and infestations) | 15 (17)
Tonsillitis (Infections and infestations) | 15 (21)
Corona virus infection (Infections and infestations) | 30 (33)
Alanine aminotransferase increased (Investigations) | 19 (26)
Aspartate aminotransferase increased (Investigations) | 13 (17)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 16 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (17)
Headache (Nervous system disorders) | 13 (16)
Psoriasis (Skin and subcutaneous tissue disorders) | 13 (16)
Hypertension (Vascular disorders) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03355573/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03355573/SAP_001.pdf